CLINICAL TRIAL: NCT07250139
Title: Comparative Study of Ziplyft Treatment vs. Traditional Blepharoplasty for Upper Eyelid Rejuvenation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osheru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25592-Osheru
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Dermatochalasis of Upper Eyelid; Ptosis, Eyelid; Blepharoplasty
Keywords: Dermatochalasis of upper eyelid, Ptosis of upper eyelid, blepharoplasty,; Ziplyft; upper eyelid surgery
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Intervention Model Description: This study will be conducted using a "split-face" design. For each participant, one eyelid will be treated with the traditional blepharoplasty method and the other with Ziplyft, allowing a direct side-by-side comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Comparing Ziplyft Device Treatment to Standard Blepharoplasty (Experimental): Ziplyft is a Class 1, 510(k) Exempt device for removing excess unwanted eyelid skin. Ziplyft will be used on one side of the participant's face to compress the excess skin prior to excess eyelid skin removal.
  Standard blepharoplasty will be performed on the fellow side of the participant's face.
  Interventions: Device: Ziplyft Device; Other: Comparator Arm: Standard Blepharoplasty

INTERVENTIONS:
Device: Ziplyft Device — Ziplyft will be used on one side of the participant's face to compress the excess skin prior to excess eyelid skin removal. Ziplyft compresses the excess skin and seals it together, no suturing is required, and the surgery incision will be closed with tissue adhesive.
Other: Comparator Arm: Standard Blepharoplasty — Standard blepharoplasty will be used on the fellow side of the participant's face. Standard blepharoplasty uses a blade, cautery to seal blood vessels, and sutures to close the incision.

SUMMARY:
This study will compare two surgery techniques used for upper eyelid (eyelift) surgery: traditional surgery and a newer method called Ziplyft (a non-powered, hand-held clamp). This study will use a "split-face" design, meaning one eyelid will be treated with the traditional surgery method and the other with Ziplyft, allowing a direct side-by-side comparison.

The objectives of the study are to compare Ziplyft treatment vs. traditional surgery by evaluating bruising, wound closure and incision, surgery case time, and subject/surgeon surveys.

DETAILED DESCRIPTION:
Blepharoplasty (upper eyelid surgery), is a procedure where excess upper eyelid skin that can interfere with peripheral vision is removed, resulting in improvement in peripheral vision and a more revitalized appearance. The amount of excess skin to be removed from each lid is marked symmetrically on both right and left sides just as it is in a standard blepharoplasty. The difference in this comparative study is that one side will be done using a blade, cautery to seal blood vessels, and sutures to close the incision which is how a standard blepharoplasty procedure is performed. On the other side, the exact same amount of tissue that was marked prior to the surgery will be removed. The fellow (second) side will use a clamp (Ziplyft) to compress the excess skin prior to removal so that there is no bleeding and therefore no need for cautery to seal blood vessels. The same amount of tissue will be removed on this second side; it will be all the marked tissue. As the clamp compresses the excess skin and seals it together, no suturing is required, and the incision can be closed with tissue adhesive which has been used for many years to close eyelid surgery incisions. Using the commercially available tissue adhesive eliminates the need for sutures to close the incision. Both right and left upper eyelids will have the same amount of tissue removed, similar to standard blepharoplasty surgery. Both sides will also have incisions; one will be closed with sutures, and the other will be closed with tissue adhesive. In summary, both right and left upper eyelids are getting a standard blepharoplasty procedure. One side is utilizing a clamp (Ziplyft) to eliminate bleeding and the need for sutures.

The surgeon will record case time for Ziplyft side and traditional blepharoplasty side. Post-op photos taken at day 3 and 7 will be used to assess ecchymosis (bruising) by a masked, independent professional (physician). Photos taken at 7 days and 1-month post-op with lids closed and lids open will be rated on incision appearance by a masked, independent professional (physician). Participant- and surgeon-reported surveys will be used to evaluate satisfaction with the Ziplyft procedure and outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed written consent prior to participation in any study-related procedures.
2. Ability, comprehension, and willingness to follow study instructions, and likely to complete all study visits.
3. Male or female adults, ≥ 35 years old at the Preoperative Visit willing to return for required follow-up visits.
4. Subjects with excess eyelid skin are eligible to undergo the procedure in the opinion of the investigator.
5. Female subjects must be 1-year postmenopausal, surgically sterilized, or, if of childbearing potential, have a negative urine pregnancy test at the Preoperative Visit. Women of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include at least one of the following: intrauterine (intrauterine device), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.

Exclusion Criteria:

1. Subjects with a current Ptosis diagnosis
2. Subjects with a history of Graves' Disease
3. Subjects with Myasthenia Gravis
4. Subjects that in the opinion of the investigator are anatomically not conducive to using devices (e.g., heavy brow, severe hollowing of the upper eyelid, history of ocular or orbital trauma).
5. Subjects that have had any previous surgery eyelid or eyebrow region.
6. Use of anticoagulation therapy, including, but not limited to Aspirin, NSAIDS, Ibuprofen within 7 days and Xarelto, Warfarin, Enoxaparin, Plavix within 3 days prior to planned study procedure.
7. Active or recent (within 3 months) tobacco user
8. Allergy to adhesive glue
9. Participation in any study of an investigational, interventional product within 30 days prior to the Preoperative Visit or at any time during the study period.
10. Pregnant or nursing females.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Compare surgical case time for Ziplyft treatment versus standard blepharoplasty | From the beginning of the surgical case until surgery has been completed
  The surgeon will record the surgical case times for Ziplyft and standard blepharoplasty. For the Ziplyft side of the participant's face the surgical case time begins when the Ziplyft device touches the patient lid and ends 1 min after adhesive is applied as that is when it has cured. For the standard blepharoplasty side of the participant's face the surgical case time begins as the blade begins its first cut and ends once ointment has been applied.
Document post-operative ecchymosis with Ziplyft and standard blepharoplasty | 3 days following surgery (±1 day) to 9 days after the surgery (± 3 days)
  Ecchymosis will be measured by post-operative photographs taken at day 3 and day 7. Photos will be rated on a 1-4 scale for ecchymosis by an independent masked observer (physician).
Measure the success of tissue adhesive (Ziplyft side) versus suture (standard blepharoplasty side) for wound closure and incision appearance. | 9 days (± 3 days) to up to 2 months (± 1 month) post-operation
  Photos taken at 9 days and 1-month post-op with lids closed and lids open will be rated on incision appearance by an independent masked observer (physician).
Assess patient reported outcomes with Ziplyft versus standard blepharoplasty | After the surgery is completed (post-operation on the day of the procedure) until 2 months (± 1 month) post operation
  Patient satisfaction questionnaires regarding comfort, satisfaction, and healing experience will be administered to the participants on the day of surgery and at 2 months post operation.
Evaluate surgeon-reported experiences with Ziplyft and standard blepharoplasty | The day of surgery until 2 months (± 1 month) post-operation
  A surgeon-reported questionnaire regarding the procedure efficiency, bleeding, and the use of cautery and suture will be administered following the surgical procedure. A second surgeon-reported questionnaire regarding the use of adhesive, bruising, swelling, scaring, and symmetry will be administered at 2-months post operation.

CONTACTS AND LOCATIONS:
Locations (1):
- New Century Ophthalmology, Oxford, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No